CLINICAL TRIAL: NCT01155960
Title: An Open Label, Balanced, Randomized,Two-Treatment, Two-Sequence, Two Period, Crossover, Single Dose Comparative Oral Bioavailability Study Of Anastrozole Tablets 1 mg (Test) Of Dr. Reddy's Laboratories Ltd., India And ARIMIDEX® Tablets 1 mg (Reference) Of Astrazeneca Pharmaceuticals LP, USA In Post Menopausal Healthy Women Subjects Under Fed Conditions.
Brief Title: Bioavailability Study of Anastrozole Tablets 1 mg of Dr.Reddy's Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Dr. Ramesh Mullangi -Director, Dr.Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BA0859094
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Bioavailability; Anastrozole; Crossover
MeSH Terms: interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arimidex (Active Comparator): Arimidex® Tablets 1 mg
  Interventions: Drug: Anastrozole
- Anastrozole (Experimental): Anastrozole Tablets 1 mg of Dr.Reddy's Laboratories Limited
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole — Anastrozole Tablets 1 mg of Dr.Reddy's Laboratories Limited
  Other Names: Arimidex® Tablets 1 mg

SUMMARY:
The purpose of this study is to compare bioavailability in healthy, post menopausal women subjects under fed conditions.

DETAILED DESCRIPTION:
Open label, balanced, randomized, two treatment, two-sequence, two periods, crossover, single dose, comparative oral bioavailability study in healthy, post menopausal women subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects should be postmenopausal healthy women who have attained complete menopause naturally or surgically and have not had menstruation for at least one year and are not on hormone replacement therapy.
2. The subjects should have Estradiol level ≤ 20 pg/ml & serum follicular stimulating hormone (FSH) level ≥ 50 mlU/ml during the screening.
3. The subjects should be screened within 21 days prior to the administration of first dose of the study drug.
4. The subjects should have a BMI between 18.5 to 26.4 (30-39 years), 18.5 to 27.8 (40-49 years), 18.5 to 28.4 (50-59 years) & 18.5 to 27.5 (60-69 years) weight in kg/ height2 in meter.
5. The subjects should be able to communicate effectively with study personnel.
6. The subjects should be able to give written informed consent to participate in the study.

Exclusion Criteria:

1. The subjects who have a history of allergic responses to Anastrozole or other related drugs.
2. The subjects who are using female hormone replacement therapies, thyroid hormone replacement therapies, or antihypertensive therapies.
3. The subjects who have significant diseases or clinically significant abnormal findings during screening, (medical history, physical examination, laboratory evaluations, ECG, X-ray & lower abdominal ultrasonography recordings).
4. The subjects who have any disease or condition which might compromise the haemopoeitic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system, diabetes, psychosis or any other body system.
5. The subjects who have a history or presence of bronchial asthma.
6. The subject who have used of enzyme-modifying drugs within 30 days prior to receiving the first dose of study medication.
7. The subjects who have history of drug dependence, recent history of alcoholism or of moderate alcohol use.
8. The subjects who are smokers, who smoke more than or equal to 10 cigarettes per day or more than or equal to 20 biddies per day or those who cannot refrain from smoking during study period.
9. The subjects with a history of difficulty with donating blood or difficulty in accessibility of veins.
10. The subjects who have donated (1 unit: 350 ml / 450 ml) blood within 90 days prior to receiving the first dose of study medication.
11. The subjects who have a positive hepatitis screen (includes subtypes A, B, C & E).
12. The subjects who have a positive test result for Human Immunodeficiency Virus (HIV) antibody and / or syphilis Rapid Plasma Reagin, Venereal Disease Research Laboratory (RPR/VDRL).
13. The subject who received an investigational product, or has participated in a drug research study within a period of 90 days prior to the first dose of the study medication administration.

Ages: 37 Years to 67 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Bioavailability based on Cmax and AUC parameters | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ronak Modi, MBBS, Principal Investigator — BA Research India Ltd.,